CLINICAL TRIAL: NCT03940027
Title: EUS-guided Celiac Plexus Neurolysis Using Ropivacaine Combined With Anhydrous Alcohol for the Treatment of Abdominal Pain in Pancreatic Cancer: a Prospective Multicenter Randomized Clinical Trial
Brief Title: EUS-guided Celiac Plexus Neurolysis for the Treatment of Abdominal Pain in Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); Shanghai Cancer Hospital, China (Other); The Third Xiangya Hospital of Central South University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, chief of the Gastroenterology, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPN
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Pancreatic Cancer
Keywords: EUS-guided CPN
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The included patients were divided into two groups (stage III and stage IV) according to tumor staging, and the patients in the two groups were randomly divided into two groups for EUS-CPN treatment with ropivacaine + anhydrous alcohol regimen and bupivacaine + anhydrous alcohol regimen
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ropivacaine (Experimental): The patients will be carried on EUS-CPN with 10ml 0.75% ropivacaine with 10ml anhydrous alcohol
  Interventions: Procedure: EUS-guided celiac plexus neurolysis
- bupivacaine (Active Comparator): The patients will be carried on EUS-CPN with 10ml 0.75% bupivacaine with 10ml anhydrous alcohol
  Interventions: Procedure: EUS-guided celiac plexus neurolysis

INTERVENTIONS:
Procedure: EUS-guided celiac plexus neurolysis — EUS-guided celiac plexus neurolysis (EUE-CPN) is an endoscopic ultrasound-guided injection of local anesthetics and neurodegenerative agents into the abdominal ganglion area through the gastric wall, so as to achieve irreversible damage of the abdominal nerve and interrupt the pain pathway of pancreatic cancer.EUS-CPN has the advantages of less trauma, higher technical success rate and lower risk of complications compared with traditional ct-guided CPN in vitro puncture.The data showed that eus-cpn was effective in the treatment of pancreatic cancer related persistent abdominal pain up to about 70%, significantly reducing the dosage of analgesics and improving the quality of life of patients with advanced pancreatic cancer.

SUMMARY:
Studies have shown that injecting local anesthetics in areas rich in blood vessels increases the risk of drug injection into blood vessels by mistake and increases the systemic absorption of drugs, which may increase the incidence of central nervous system and cardiovascular system toxic events caused by local anesthetics.EUS-CPN-related complications have not been clearly associated with local anesthetic adverse events.However, EUS-CPN local anesthetic injection area is located around the beginning of the abdominal trunk with abundant large and small blood vessels. The choice of local anesthetics with higher safety than bupivacaine, such as ropivacaine, is of great significance to ensure the safety of eus-cpn, especially for eus-cpn beginners.At present, there are no reports on the application of ropivacaine in eus-cpn.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-75;
2. Athologically confirmed as pancreatic cancer and clinically evaluated as advanced and unresectable;
3. The visual analogue scale (VAS) for pain ≥ 4；
4. Never received treatment for peritoneal plexus lesion or block；
5. Voluntary signing of written informed consent

Exclusion Criteria:

1. Women during pregnancy；
2. Cannot or refuses to sign the informed consent；
3. Blood clotting disorder（PLT <50 × 103/μL, INR > 1.5）；
4. Celiac infection；
5. Severe esophageal or gastric varices and ulcers which may affect operation;
6. The anatomical variation of the abdominal trunk abdominal aorta and could not be accurately located;
7. Alcohol allergy
8. Severe cardiopulmonary dysfunction and inability to tolerate the risk of intravenous anesthesia;
9. History of mental illness;
10. Patients with other chronic and acute diseases with unstable conditions that are expected to affect the efficacy evaluation and completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The effective rate of abdominal pain relief | 2 weeks
  Preoperative and postoperative pain scores of the patients will be compared to estimate the effective rate of abdominal pain relief.
the incidence of serious complications | 2 weeks
  Complications like perforation, infection, pancreatitis, hemorrhage and local anesthetic complications (epilepsy, arrhythmia), etc.

SECONDARY OUTCOMES:
Improvement of quality of life | 1 month, 3 months, 6 months and 1 year
  Preoperative and postoperative quality of life questionnaire of the patients will be compared to estimate the improvement of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-shen Li, Ph.D., Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No